CLINICAL TRIAL: NCT02826109
Title: The Efficacy of Cyanoacrylate (PeriAcryl®90 HV) in Its Adhesive Post-Operative Properties on Periodontal Wound Healing and Patient Discomfort After Non-Surgical Periodontal Treatment: A Pilot Randomized Clinical Trial
Brief Title: The Efficacy of Cyanoacrylate Adhesive (PeriAcryl®90 HV) in Periodontal Wound Healing
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H15-03277
Record Dates: First submitted 2016-06-06; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Periodontal Disease; Tissue Adhesive; Dental Scaling; Wound Healing; Oral Surgical Procedures; Pain
MeSH Terms: conditions — Periodontal Diseases; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional: Cyanoacrylate Application (Experimental): Application of cyanoacrylate adhesive to one quadrant of mouth
  Interventions: Device: PeriAcryl®90 HV
- Control: Absence of Cyanoacrylate Application (No Intervention): No application of cyanoacrylate adhesive to the other quadrant of mouth

INTERVENTIONS:
Device: PeriAcryl®90 HV
  Arms: Interventional: Cyanoacrylate Application

SUMMARY:
Periodontal disease is a gum infection caused by plaque on teeth containing both bacteria and calculus (hard) deposits. These need to be removed on a regular basis to maintain gum health and to prevent teeth weakening. A routine cleaning procedure, scaling/root planing, is accompanied with post-operative soft tissue tenderness and teeth sensitivity making oral hygiene maintenance difficult during wound healing. The need for novel therapeutic approaches, such as cyanoacrylate adhesives, has been identified. It has been hypothesized that its application may provide comfort and assist patients with their daily oral self-care procedures following teeth cleaning.

DETAILED DESCRIPTION:
Hypothesis: The supra-gingival marginal application of cyanoacrylate adhesive will promote periodontal wound healing and prevent the increase of sensitivity of hard (teeth) and soft (gingiva) tissues following non-surgical periodontal therapy (NSPT).

This pilot study involves a small number of participants, and while it is not designed to prove causation, it will evaluate safety and efficacy. If clinical results are positive, these data may be used to determine sample and power needs for larger studies.

With enhanced post-operative comfort, the patient's ability to disrupt biofilm and maintain optimal daily oral self-care can be achieved. Biofilm disruption is paramount to achieving periodontal health. Specifically, the adjunctive placement of an adhesive dressing may reduce biofilm accumulation that is associated with periodontal inflammation. This novel application could improve the patient's oral and thus overall health.

The present pilot trial aims to explore the therapeutic effectiveness of a cyanoacrylate adhesive (PeriAcryl®90 HV) in reducing patient-reported outcomes related to discomfort and sensitivity post NSPT, examine their potential positive effects on periodontal wound healing as well as recording any potential side-effects that may have been experienced by the patients.

ELIGIBILITY:
Inclusion Criteria:

The potential subjects must:

* Be capable of giving informed consent and 19 years of age or older
* Have a minimum of 18 teeth and at least 4 measurement sites with pocket depth at least 5.0 mm with bleeding on probing in at least 2 different quadrants
* Be able to understand and communicate in English, as the study cannot fund a certified interpreter
* Be willing and able to return for treatment and evaluation throughout the course of this study.

Exclusion Criteria:

Potential subjects must not:

* Have had any antibiotics in the last month
* Be pregnant, nursing or plan to become pregnant over the course of the trial
* Have an active smoking history (tobacco or otherwise)
* Have sites with overt abscess, active caries or crown/root fractures
* Have known adverse reactions or allergies to cyanoacrylates or formaldehyde
* Have any other significant disease or take medication(s) that, in the opinion of the investigator, may interfere with the evaluation of safety or efficacy of cyanoacrylate and overall compliance.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-05 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Prevention of increased post-operative discomfort post placement of cyanoacrylate adhesive measured by Visual Analogue Scale | after 6-8 weeks
Change in clinical attachment levels (CAL) after NSPT with adjunctive placement of cyanoacrylate adhesive | after 6-8 weeks
Prevention of increased hypersensitivity (hard and soft dental tissues) after NSPT post placement of cyanoacrylate adhesive measured by Visual Analogue Scale | after 6-8 weeks
Continued relief post placement of cyanoacrylate adhesive measured by Visual Analogue Scale | after 6-8 weeks

SECONDARY OUTCOMES:
Subjects' compliance to having the cyanoacrylate adhesive post-operatively by interview and tabulation of patient-reported outcomes | after 6-8 weeks
Number of adverse reactions to the placement of cyanoacrylate adhesive at the supra-gingival margin | after 6-8 weeks
Change in probing pocket depth (PD) | after 6-8 weeks
Change in bleeding on probing (BOP) | after 6-8 weeks
Change in plaque scores | after 6-8 weeks
Subjects' perception of having the cyanoacrylate adhesive post-operatively by interview and tabulation of patient-reported outcomes | after 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Penny Hatzimanolakis, DipDH, BDSc, MSc, RDH, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada